CLINICAL TRIAL: NCT01429467
Title: Improving Glucose Variability in Type 1 Diabetes and Its Effect on the Underlying Homeostatic Metabolic Pathways of Angiogenesis
Brief Title: Glucose Variability in Type 1 Diabetes and Its Effect on Factors That Influence New Vessel Formation
Acronym: INDIGO 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Anthony Tasker, SCREDS Lecturer, University of Dundee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AT/V01/010911
Record Dates: First submitted 2011-09-01; First posted 2011-09-07 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes
Keywords: Glucose Variability; Continuous Glucose Monitoring; Hypoxia-inducible Factor (HIF); Vascular Endothelial Growth Factor (VEGF); Erythropoietin; Cortisol
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Continuous Glucose Monitoring (CGM) (Other): 10 participants from phase 1 will undergo 6 weeks of CGM with telemedicine support at weeks 1,3 + 5. After this period HIF, Erythropoietin, VEGf and cortisol will again be measured and compared with the subjects glucose variability.
  Interventions: Device: Continuous Glucose Monitor (CGM) and Telemedicine (Enlite Guardian real-time system Medtronic®)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) and Telemedicine (Enlite Guardian real-time system Medtronic®) — Phase 2 patients will receive 6 weeks of CGM (Enlite Guardian real-time system- Medtronic®). Optimisation of glycaemic control will be through a telemedicine system to deliver a standardised protocol to instruct changes in pump settings and insulin delivery rate. This has been devised in our department and used successfully in a clinical trial comparing MDI v. CSII in young people, sponsored by Diabetes UK. 2008-2010). Subjects will be contacted at 1, 3 and 5 weeks after starting the CGM
  Other Names: Enlite Guardian real-time system Medtronic®

SUMMARY:
The aim of the study is to see how glycaemic control and glycaemic variability affect levels of HIF, VEGF, erythropoietin and cortisol in Paediatric Type 1 diabetics on insulin pump therapy.

DETAILED DESCRIPTION:
The study will have two parts. The first phase will look at all current paediatric type 1 diabetics in Tayside on continuous subcutaneous insulin pump therapy and measure their levels of Hypoxia-Inducible Factor (HIF), Vascular Endothelial Growth Factor (VEGF), erythropoietin and cortisol. This will help answer the question; Does glucose control (as expressed by HbA1c ) effect levels of HIF, VEGF, erythropoietin and cortisol? To our knowledge this will be the first human study comparing how HIF, VEGF, erythropoietin and cortisol are affected by glucose control

The second phase of the trial will chose 10 patients on insulin pump therapy and using a continuous glucose monitor (CGM), monitor their glucose variability over a period of 6 weeks. After this period their levels of HIF, VEGF, erythropoietin and cortisol will again be measured. This will help answer the question of whether there is a relationship between glucose variability and levels of HIF, VEGF, erythropoietin and cortisol. As we know that these factors are stimulated by episodes of hypo and hyperglycaemia, it is hypothesised that these factors will be lower in participants that demonstrate reduced glucose variability. It will be the first study to give detailed information on the relationship between HIF, VEGF, erythropoietin and cortisol and glucose variability.

By using telemedicine sessions during weeks 1, 3 and 5 of the participants wearing CGM we will aim to improve the participant's glucose variability. This will help give further information about glucose variability and the above factors as well as giving further evidence for the use of telemedicine and CGM to improve glycaemic control in adolescent diabetics.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 inclusion:

* Patients with Type 1 Diabetes
* On insulin pump therapy.
* Aged 5 years to 18 years.

Phase 2 inclusion:

* Patents with Type 1 Diabetes
* Diabetes diagnosis for 1 year
* On insulin pump therapy for minimum of six months
* Access to a computer with internet access and telephone
* Agree to wear CGM for 6 weeks
* Aged 12 years to 18 years

Exclusion Criteria:

* Patients not on pump therapy
* Patient less than 5 years and greater than 18 years
* Phase 2 patients been on pump therapy for less than 6 months
* Phase 2 patients without access to internet and telephone.
* Phase 2 patients less than 12 years and greater than 18 years
* Patients who do not have a good understanding of English

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Correlation of HbA1c and level of Hypoxia-inducible Factor | Baseline
  This will look at all the results from Phase 1 participants and see if their is a correlation between participants HbA1c and their level of Hypoxia-inducible factor.
Correlation of HbA1c and level of Vascular Endothelial Growth Factor | Baseline
  This will look at all the results from Phase 1 participants and see if their is a correlation between participants HbA1c and their level of Vascular Endothelial Growth Factor.
Correlation of HbA1c and level of Erythropoietin | Baseline
  This will look at all the results from Phase 1 participants and see if their is a correlation between participants HbA1c and their level of Erythropoietin.
Correlation of HbA1c and level of cortisol | Baseline
  This will look at all the results from Phase 1 participants and see if their is a correlation between participants HbA1c and their level of Cortisol.

SECONDARY OUTCOMES:
Change in Mean Area of Glucose Excursion (MAGE) following CGM | 6 weeks
  The Mean Area of Glucose Excursion (MAGE) will be calculated for all phase 2 particpants from the CGM data in the first 3 days and last 3 days of the 6 week CGM period. These will then be compared to see if there is a statistical difference between MAGE after CGM intervention.
Change in levels of Hypoxia-inducible factor following CGM | 6 weeks
  Levels of Hypoxia-inducible factor will be measured in phase 2 participants post CGM and compared with baseline Hypoxia-inducible factor taken in phase 1 to see if there is a statistical difference.
Change in levels of Vascular Endothelial Growth Factor following CGM | 6 weeks
  Levels of Vascular Endothelial Growth Factor will be measured in phase 2 participants post CGM and compared with baseline Vascular Endothelial Growth Factor taken in phase 1 to see if there is a statistical difference.
Change in levels of erythropoietin following CGM | 6 weeks
  Levels of Erythropoietin will be measured in phase 2 participants post CGM and compared with baseline Erythropoietin taken in phase 1 to see if there is a statistical difference.
Change in levels of cortisol following CGM | 6 weeks
  Levels of Cortisol will be measured in phase 2 participants post CGM and compared with baseline Cortisol taken in phase 1 to see if there is a statistical difference.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony PB Tasker, MBChB, Principal Investigator — University of Dundee
Locations (1):
- University Of Dundee, Dundee, Angus, United Kingdom